CLINICAL TRIAL: NCT01424930
Title: An Open-Label Study to Determine the Short-Term Safety of Continuous Dosing of Abiraterone Acetate and Prednisone in Modified Fasting and Fed States to Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study to Determine the Short-Term Safety of Continuous Dosing of Abiraterone Acetate and Prednisone in Modified Fasting and Fed States to Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018715; 212082PCR2008 (Other: Janssen-Ortho, Canada)
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Neoplasms; Prostate Cancer
Keywords: Metastatic castration-resistant prostate cancer; CRPC; Abiraterone Acetate; Prednisone; Food Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abiraterone+prednisone (low-fat meal) (Experimental): Participants will receive abiraterone acetate at a starting dose of 1,000 milligram (mg) once daily for 7 days post 30-minutes of a standardized low-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14. Prednisone will be administered as 5 mg oral tablet twice daily during Cycle 1 Day 8 to Cycle 1 Day 14.
  Interventions: Drug: Abiraterone; Drug: Prednisone
- Abiraterone+prednisone (high-fat meal) (Experimental): Participants will receive abiraterone acetate at a starting dose of 1,000 mg once daily for 7 days post 30-minutes of a standardized high-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14. Prednisone will be administered as 5 mg oral tablet twice daily during Cycle 1 Day 8 to Cycle 1 Day 14.
  Interventions: Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone — Participants will receive abiraterone acetate at a starting dose of 1,000 mg once daily for 7 days post 30-minutes of a standardized low-fat meal and high-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14.
Drug: Prednisone — Prednisone will be administered as 5 mg oral tablet twice daily during Cycle 1 Day 8 to Cycle 1 Day 14.

SUMMARY:
The purpose of this study is to establish the safety profile of oral (by mouth) abiraterone acetate and oral prednisone following short-term administration after standardized low-fat or high-fat meals to patients with metastatic (spreading) castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a multicenter, open-label study of 24 (up to a total of 28) men to assess the short-term safety of oral abiraterone acetate 1 g and oral prednisone 5 mg twice daily administered in the modified fasted state and after meals of various fat contents. All patients will take daily abiraterone acetate for the first 7 days in the modified fasted state (no food for 2 hours before and 1 hour after the dose). In Cohort 1, up to 6 evaluable patients will take abiraterone acetate daily for 7 days after a standardized low-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14; or, in Cohort 2, up to 6 evaluable patients will take abiraterone acetate daily for 7 days after a standardized high-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14. All patients will then continue to take abiraterone acetate daily in the modified fasted state starting on Cycle 1 Day 15 until disease progression. Toxicity related to dosing after the low-fat or high-fat meals is defined as Grade 3 or higher AEs of special interest; or Grade 3 or higher serious adverse events (SAEs) that occur during the food safety evaluation period. Cohort 2 may be expanded to a total of 18 evaluable patients if deemed to be safe. Decisions regarding the escalation of cohort or expansion of cohorts will be made by a study evaluation team. Pharmacokinetic evaluation for each cohort will be performed on Cycle 1 Days 7 and 14 at predose and multiple timepoints postdose over 24 hours; Cycle 1 Days 8 and 11 at 2 hours following abiraterone acetate dose administration. Abiraterone acetate, 1 g (four 250-mg tablets) orally (taken by mouth) once daily. Patients may take abiraterone acetate until progression of clinical disease. Prednisone, 5 mg, orally, twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Metastatic disease documented by bone, computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Surgical or medical castration with testosterone less than 50 ng/dL (< 2.0 nM)
* Prostate-specific antigen (PSA) or radiographic progression documented by assessments specified in study protocol
* Platelets >100,000/µl
* Hemoglobin >=9.0 g/dL
* Liver function tests (LFTs): Serum bilirubin < 1.5 x ULN; AST or ALT < 2.5 x ULN; Eastern Cooperative Oncology Group (ECOG) status score of <=2

Exclusion Criteria:

* Small cell carcinoma of the prostate
* Known brain metastasis, chronic liver disease with elevated LFTs
* Prior cytotoxic chemotherapy for metastatic prostate cancer
* Treatment of prostate cancer within 30 days of Day 1 Cycle 1 with surgery, radiation, chemotherapy or immunotherapy
* Use of investigational drug within 30 days of Day 1 Cycle 1 or current enrollment in an investigational drug or device study
* Recent history of ischemic heart disease, Electrocardiogram (ECG) abnormalities or atrial fibrillation
* Active infection or other medical condition that would make prednisone (corticosteroid) use contraindicated
* Chronic medical condition requiring a higher dose of corticosteroid than prednisone 5 mg twice daily

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho, Canada Clinical Trial, Study Director — Janssen-Ortho Inc., Canada
Locations (2):
- Canada (2):
  - Edmonton, Alberta
  - Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 29 September 2011 to 29 May 2013. Participants were recruited at 2 study centers in Canada.
Groups:
- Abiraterone+Prednisone (Low-fat Meal): Participants received abiraterone acetate at a starting dose of 1,000 milligram (mg) once daily for 7 days post 30-minutes of a standardized low-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14. Prednisone was administered as 5 mg oral tablet twice daily during Cycle 1 Day 8 to Cycle 1 Day 14.
- Abiraterone+Prednisone (High-fat Meal): Participants received abiraterone acetate at a starting dose of 1,000 mg once daily for 7 days post 30-minutes of a standardized high-fat meal from Cycle 1 Day 8 to Cycle 1 Day 14. Prednisone was administered as 5 mg oral tablet twice daily during Cycle 1 Day 8 to Cycle 1 Day 14
Period: Overall Study
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal)
Started | 7 | 18
Completed Food Safety Evaluation | 6 | 18
Completed | 3 | 4
Not Completed | 4 | 14
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Progressive Disease | 3 | 6
Not completed — Screen Failure | 0 | 1
Not completed — Reason not specified | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal) | Total
Number analyzed (Participants) | 7 | 18 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (11.01) | 69.1 (7.26) | 70.8 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 18 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Events (AEs) of Special Interest or Grade 3 or Higher Serious AEs Due to Study Medication
Description: AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Events with Grade 3 or higher (3=Severe; 4=life-threatening; 5=fatal) are events that significantly interrupt usual daily activity, require systemic drug therapy/other treatment and are, in many situations, considered unacceptable or intolerable events.
Time Frame: Postdose on Cycle 1 Day 8 to predose on Cycle 2 Day 1
Population: Safety population: Participants who received at least 1 dose of study medication and contributed any safety data after the start of study treatment.
Measure: Number; unit: Participants
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal)
Number analyzed (Participants) | 6 | 18
Participants | 0 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Abiraterone
Description: The table below shows mean Cmax of Abiraterone. The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Time Frame: Day 7 and Day 14
Population: Participants who received at least 1 dose of study medication and were included in the pharmacokinetics analysis.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal)
Number analyzed (Participants) | 7 | 18
ng/mL
  Day 7 | 218 (168) | 196 (234)
  Day 14 | 265 (229) | 342 (289)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Abiraterone
Description: The table below shows median Tmax of Abiraterone. The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time Frame: Day 7 and Day 14
Population: Participants who received at least 1 dose of study medication and were included in the pharmacokinetics analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal)
Number analyzed (Participants) | 7 | 18
hours
  Day 7 | 2 (1.0 - 8.1) [1.0 to 8.1] | 2 (0.5 - 6.0) [0.5 to 6.0]
  Day 14 | 2.5 (1.0 - 3.0) [1.0 to 3.0] | 4.0 (3.0 - 10.0) [3.0 to 10.0]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration to 24 Hours After Dosing (AUC24h)
Description: The table below shows mean AUC24h. The Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: Day 7 and Day 14
Population: Participants who received at least 1 dose of study medication and were included in the pharmacokinetics analysis.
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal)
Number analyzed (Participants) | 7 | 18
ng*h/mL
  Day 7 | 1271 (1279) | 973 (667)
  Day 14 | 1264 (963) | 1992 (720)

ADVERSE EVENTS:
Arm/Group | Abiraterone+Prednisone (Low-fat Meal) | Abiraterone+Prednisone (High-fat Meal)
Serious Adverse Events (participants affected / at risk) | 4/7 | 4/18
Other Adverse Events (participants affected / at risk) | 7/7 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone+Prednisone (Low-fat Meal) (N=7) | Abiraterone+Prednisone (High-fat Meal) (N=18)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone+Prednisone (Low-fat Meal) (N=7) | Abiraterone+Prednisone (High-fat Meal) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1
Blindness Transient (Eye disorders) | 0 | 1
Eye Swelling (Eye disorders) | 1 | 1
Ocular Hyperaemia (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0
Visual Impairment (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Dry Mouth (Gastrointestinal disorders) | 1 | 2
Faecal Incontinence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 2
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 7
Oral Discharge (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 4
Chills (General disorders) | 1 | 1
Facial Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 11
Gait Disturbance (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 3
Oedema Peripheral (General disorders) | 4 | 6
Pyrexia (General disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Cystitis (Infections and infestations) | 0 | 3
Gastroenteritis Viral (Infections and infestations) | 1 | 1
Herpes Zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral Herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
Weight Increased (Investigations) | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis of Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 1
Disturbance in Attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 0 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 2 | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1
Sinus Headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
"hallucination (Psychiatric disorders) | 0 | 1
Abnormal Dreams (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Mental Disorder (Psychiatric disorders) | 0 | 1
Bladder Spasm (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Loss of Bladder Sensation (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 2
Urinary Hesitation (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 2
Breast Pain (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flush (Vascular disorders) | 2 | 5
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 2
Peripheral Coldness (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days